CLINICAL TRIAL: NCT00029783
Title: Efficacy of Distant Healing in Glioblastoma Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: R01AT000644-03 (NIH); NCT00058500 (obsolete NCT alias)
Record Dates: First submitted 2002-01-23; First posted 2002-01-24 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; Brain tumor; Distant healing; Distance healing
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

INTERVENTIONS:
Procedure: Distant Healing

SUMMARY:
This study will assess whether distant healing effects survival time and loss of function for glioblastoma patients.

DETAILED DESCRIPTION:
Prayer, energy healing, and spiritual healing are widely used for all degrees of illness.

Eisenberg (1998) reported that more that 26% of his survey sample used "energy healing" within the last year. Most of these practitioners believe that their inner intentions result in the benefits, either through the agency of love, energy, or a Higher Power (Benor 1992). However, the conventional community attributes benefits from these interventions to the patient's hope, expectation, or experience of support from a practitioner (Benson 1996). The proposed study is a double-blind randomized controlled clinical trial of "distant healing intentionality." Distant Healing (DH) is defined as a "mental intention on behalf of one person, to benefit another at a distance." This study will assess whether DH effects survival time and loss of function for glioblastoma patients under conditions where hope and expectation are controlled. The study will include approximately 150 patients who have rapidly progressing glioblastoma and are beginning radiotherapy. Patients will be photographed and assessed for quality of life, psychological status, and physical symptoms as well as health habits and attitude toward DH. After stratification by age and functional status (Karnofsky score), patients will be randomly assigned to either standard treatment with or without DH. Healers from diverse schools and backgrounds from communities across the United States will be assigned to patients by rotation, so that each patient in the DH group will be treated for two weeks by 10 different healers over the 20 week intervention. Experienced healers will have photographs of subjects and send "mental intention for health and well being" to subjects for one hour daily, three times per week. The healing intervention will be performed at a distance, and patients and healers will never meet, nor will patients know their group assignment. The study findings will provide the basis for developing a larger study, definitive trial.

ELIGIBILITY:
Inclusion:

* Histologically confirmed diagnosis of glioblastoma based on open resection.
* Patient is within five weeks of diagnosis confirmed by pathology report.

Exclusion:

* Non-English speaking.
* Inability or unwillingness to fill out questionnaires.
* History of other cancers within the last 2 years (except superficial basal cell, squamous cell carcinoma of the skin), or other concurrent life-threatening conditions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2000-09; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Freinkel, MD, Principal Investigator — California Pacific Medical Center Research Institute
Locations (1):
- California Pacific Medical Center Research Institute, San Francisco, California, United States